CLINICAL TRIAL: NCT01980199
Title: Phase II Proof of Concept Trial to Determine Efficacy of Fexinidazole in Visceral Leishmaniasis Patients in Sudan
Brief Title: Trial to Determine Efficacy of Fexinidazole in Visceral Leihmaniasis Patients in Sudan
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEXI VL 001
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2014-07

CONDITIONS: Visceral Leishmaniasis
Keywords: visceral leishmaniasis; fexinidazole; adults; proof of concept; efficacy; safety; pharmacokinetic; pharmacodynamic
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — fexinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fexinidazole (Experimental): 600mg tablets
  3 tablets once a day for 4 days continued by 2 tablets once a day for 6 days
  Interventions: Drug: Fexinidazole

INTERVENTIONS:
Drug: Fexinidazole — 600 mg tablets given orally, after the main daily meal
  * at the daily dose of 1800 mg (3 tablets) once a day for 4 days
  * continued by 1200mg (2 tablets)once a day for 6 days

SUMMARY:
This study is designed to determine the efficacy of Fexinidazole as an oral treatment in Visceral Leishmanisasis sudanese adults patients.

The results of this proof of concept study will allow to make a decision on whether to proceed with clinical development of Fexinidazole for visceral leishmaniasis.

DETAILED DESCRIPTION:
Visceral Leishmaniasis (VL) is a neglected disease and it is fatal if left untreated.

Until recently the first line treatment in East Africa was 30 days of Sodium Stibogluconate which can be cardiotoxic. Since 2010 WHO recommended Sodium Stibogluconate and Paromomycin for 17 days which is a shorter treatment but there remains the toxicity associated with these drugs. The second line treatment is Ambisome given as 6-10 intravenous infusions, whilst this has a better safety profile than other VL regimens it is expensive.

So there is an urgent need for short course oral treatment for VL particularly in the East African region.

Fexinidazole is a 2 substituted 5-nitroimidazole formulated for oral administration. Fexinidazole through its metabolites has demonstrated potent activity againts L. donovani intracellular amastigotes in vitro and in vivo in a visceral leishmaniasis mouse model.

The dose selected for this study (1800 mg/1200 mg for 4/6 days) has been based on the dose selected for a phase II trial on Human African Trypasonomiasis. It is albeit well tolerated and is one dose level below the maximum tolerated dose level established in phase I.

The trial is designed and will be analysed according to a sequential method known as the triangular test, using day 28 data. This sequential design allows for repeated interim analysis (every 10 patients). The null hypothesis is that the proportion cured is less than or equal to 75%. The primary endpoint is initial cure at day 28. The primary population for interim analyses and interim decision making will be the per protocol population.In the final analysis of cumulative patient data, Intention to Treat and Per Protocol Population analyses will be conducted.

The conventional 6 months (day 210) follow up outcome is still an important secondary endpointfor the final decision on whether to proceed with clinical development of Fexinidazole for VL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical signs and symptoms of primary VL (fever for at least 2 weeks, splenomegaly) and diagnosis confirmed by visualization of parasites in tissue samples (lymph node, bone marrow) on microscopy.
* Patients aged between 15 and 60 years (inclusive) who are able to comply with the protocol.
* Patients for whom written informed consent has been signed by the patients themselves (if aged 18 years and over) or by parents(s) or legal guardian for patients under 18 years of age together with the patients assent.
* HIV negative status

Exclusion Criteria:

* Patients who have previously been diagnosed with VL and received anti-leishmanial treatment (ie relapse)
* Patients with BMI <16 kg/m2
* Patients with contra-indication (known hypersensitivity) to other imidazoles (e.g. ketaconazole)
* Patients suffering from a concomitant severe underlying disease (cardiac, renal, hepatic) including hepatitis B, para kala-azar dermal leishmaniasis and tuberculosis
* Patient with clinically significant ECG findings or QTcF≥ 450 msec in 2 successive ECGs
* Major surgical intervention 4 weeks prior to enrollment.
* Patients who are pregnant or lactating.
* Female patients of child bearing age who do not agree to use an acceptable method of contraception
* Patients with haemoglobin < 5g/dl.
* Patients with platelets < 40,000/mm³.
* Patients with liver function (ALT and AST) tests of more than 2 times the upper limit of the normal range.
* Patients with serum creatinine above the normal range for age and gender.
* Patients with serum potassium (K+) above the normal range
* Patients with Bilirubin more than 1.5 times the upper limit of the normal range

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Initial cure | Day 28
  Proportion of patients with an abscence of parasites in tissue aspirate and no rescue treatment administered up to and including day 28

SECONDARY OUTCOMES:
Final cure | Day 210
  Proportion of patients initially cured at day 28 (or day 56 for slow responders) with no further signs or symptoms of visceral leishmaniasis and no requirement for rescue medication during follow-up phase up to and including the day 210

OTHER OUTCOMES:
Safety endpoint | From first dose of trial medication to day 56 for non serious AEs and to day 210 for SAEs
  Proportion of patients with SAE and/or AEs leading to treatment discontinuation
Safety endpoint | From first dose of trial medication to day 56
  Proportion of patients experiencing at least one non-serious treatment emergent AE
Pharmacokinetic assessment | From day 1 to day 12
  Whole blood concentration of Fexinidazole and metabolites (sulfone and sulfoxide) in an intensive cohort of 10 patients (18 sampling time points) and in a regular cohort for all other patients (6 sampling time points)
Pharmacodynamic assessment | Screening, D1, D3, D5, D8, D11, D14, D28, D56, D210
  Parasite load in blood and bone marrow (if remainder of bone marrow aspirate sample) to follow parasite clearance rate

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Musa, MD PhD, Principal Investigator — Director, Institute of Endemic Diseases, University of Khartoum Associate Professor, Head, Department of Clinical Pathology & Immunology; E. AG Khalil, Prof. MD, Principal Investigator — Institute of Endemic Diseases (IED), University of Khartoum
Locations (1):
- Doka Hospital, Doka, Al Qaḑārif, Sudan